CLINICAL TRIAL: NCT06630767
Title: Enhanced Recovery After Surgery Program Versus Conventional Care for Laparoscopic Common Bile Duct Exploration: A Randomized Controlled Trial
Brief Title: Enhanced Recovery After Surgery Program Versus Conventional Care for Laparoscopic Common Bile Duct Exploration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed Omar, MD, Professor Mohammed Ahmed Omar, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SVU/MED/SUR011/11/24/4/612
Record Dates: First submitted 2024-09-27; First posted 2024-10-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Choledocholithiasis
Keywords: enhanced recovery after surgery; laparoscopic common bile duct exploration
MeSH Terms: conditions — Choledocholithiasis | interventions — Enhanced Recovery After Surgery; Congresses as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS-LCBDE (Experimental): Patients subjected to enhanced recovery after surgery care for laparoscopic common bile duct exploration
  Interventions: Procedure: ERAS
- C-LCBDE (Active Comparator): Patients subjected to conventional care for laparoscopic common bile duct exploration
  Interventions: Procedure: Conventional

INTERVENTIONS:
Procedure: ERAS — Enhanced recovery after surgery (ERAS) programs are a combination of evidenced-based perioperative care approaches that work synergistically to improve recovery after surgery. The core elements of ERAS protocols are preoperative advice, optimization of diet, systematic analgesic and anesthetic regimes, and early mobilization.
  Other Names: Enhanced recovery after surgery
  Arms: ERAS-LCBDE
Procedure: Conventional — Conventional care for patients subjected for laparoscopic common bile duct exploration
  Arms: C-LCBDE

SUMMARY:
Laparoscopic common bile duct exploration (LCBDE) is a minimally invasive procedure to treat common bile duct stones (CBDS). Perioperative anxiety, hunger, thirst, fatigue, pain, nausea, and vomiting can influence a patient's recovery after surgery and prolong the in-hospital stay. Enhanced Recovery After Surgery (ERAS) is a modern concept that aims to improve perioperative patient care by implementing an evidence-based, patient-centered team approach. However, few reports focused on the safety and efficacy of the ERAS program in LCBDE. Therefore, this paper aims to compare the outcome of the ERAS program and conventional (C) care for patients undergoing LCBDE

DETAILED DESCRIPTION:
All patients undergoing surgery prefer to stay at the hospital for a shorter period and resume work as early as possible. The post-operative recovery and rehabilitation are influenced by numerous surgical factors such as inadequate pain management and postoperative complications, and non-surgical factors such as anxiety and stress, reduced physical activity, and unintended prolonged fasting due to improper scheduling.

Carefully planned perioperative care is approved to shorten the rehabilitation period and accelerate the recovery by preserving preoperative organ function, reducing the depth of intraoperative stress reaction, and minimizing postoperative complications, through many parameters such as emotional support, pharmacological prophylaxis, wound anesthesia, PONV prophylaxis, low-pressure pneumoperitoneum, and restricted use of surgical drains and infusions contributing to medical and economic benefit in healthcare. Two techniques are believed to improve post-operative recovery and rehabilitation; the first is the minimally invasive surgery and the second is the enhanced recovery after surgery (ERAS) program.

Laparoscopic common bile duct exploration (LCBDE) is one of the recent minimally invasive maneuvers to treat common bile duct stones (CBDS) that may be combined with laparoscopic cholecystectomy for gallbladder stones as a one-stage procedure with the advantage of minor trauma and bleeding, low postoperative complication and pain, quick recovery, and shorter hospital stay. On the contrary, It has various complications due to pneumoperitoneum and positioning including changes in cardiac output and blood pressure, decreased lung volumes, basal atelectasis, increased intrapulmonary shunting, raised airway pressures, acute postoperative pain, and postoperative nausea and vomiting (PONV).

Enhanced recovery after surgery (ERAS) programs are a recent combination of evidenced-based perioperative care approaches that work synergistically to improve recovery after surgery. The underlying mechanism of ERAS protocols is thought to be an attenuation of the peri-operative stress response and early gut function. The core elements of ERAS protocols are preoperative advice, optimization of diet, systematic analgesic and anesthetic regimes, and early mobilization. It facilitates early mobilization and nutrition by controlling pain and dyspepsia, therefore reducing the postoperative length of stay, and allowing patients to return to their usual lifestyle as promptly as possible.

Although ERAS programs have become more popular over the past decade and the Association of Surgeons of Great Britain and Ireland, and ERAS society guidelines have recommended 23 guidelines for different surgical fields, it remains controversial and conflicts with the traditional doctrine for surgery. It therefore has been slow to be implemented so far. Also, no ERAS program for LCBDE was offered till now. Therefore, this study aimed to compare the efficacy and safety of ERAS versus conventional care in LCBDE.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CBDS
* American Society of Anesthesiologists (ASA) scores of I - II
* Age 20-70 years

Exclusion Criteria:

* Severe cholangitis
* Severe pancreatitis
* Mirizzi syndrome
* Perforated gallbladder
* Biliary peritonitis
* Intrahepatic stones
* Hepatobiliary malignancy
* Pregnancy
* Conversion to open surgery
* Previous upper abdominal surgery

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Lenghth of hospital stay | 1 - 30 days
  The duration from the surgery to discharge

SECONDARY OUTCOMES:
Postoperative complications | 1 - 30 days
  the number of complications within 30 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Marwa N Alansary, Lecturer, Study Director — South Valley University; Mohammed A Omar, Professor, Principal Investigator — South Valley University
Locations (2):
- Egypt (2):
  - South Valley University, Luxor
  - South Valley University, Qina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Use of Enhanced Recovery After Surgery (ERAS) in Laparoscopic Cholecystectomy (LC) Combined with Laparoscopic Common Bile Duct Exploration (LCBDE): A Cohort Study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7510172/